CLINICAL TRIAL: NCT00895258
Title: Cognitive Training to Improve Work Outcomes in Severe Mental Illness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, ETwamley, Associate Professor of Psychiatry, UCSD, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH080150 (NIH); R01MH080150 (NIH); DSIR 82-SEDX
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Schizophrenia; Bipolar Disorder; Depression
Keywords: Schizoaffective Disorder; Major Depressive Disorder; Supported Employment; Work; Rehabilitation; Severe Mental Illness; Cognitive Training; Cognitive Rehabilitation; Cognitive Remediation
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Depression; Psychotic Disorders; Depressive Disorder, Major; Mental Disorders | interventions — Palliative Care; Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IPS-CT (Experimental): Participants will receive individual placement and support (IPS) plus cognitive training (CT).
  Interventions: Behavioral: Individual placement and support plus cognitive training (IPS-CT)
- IPS-ES (Active Comparator): Participants will receive individual placement and support (IPS) plus enhanced support (ES).
  Interventions: Behavioral: Individual placement and support plus enhanced support (IPS-ES)

INTERVENTIONS:
Behavioral: Individual placement and support plus cognitive training (IPS-CT) — One IPS plus one CT session each week for 12 weeks
  Arms: IPS-CT
Behavioral: Individual placement and support plus enhanced support (IPS-ES) — One IPS plus one ES session each week for 12 weeks
  Arms: IPS-ES

SUMMARY:
This study will compare the efficacy of two types of supportive treatments for a program called Individual Placement and Support, which helps people with severe mental illnesses find and keep jobs.

DETAILED DESCRIPTION:
Unemployment in people with severe mental illnesses (SMIs), such as schizophrenia, bipolar disorder, and major depressive disorder, has both economic and health-related costs. Unemployed people with SMIs often report an improved quality of life after finding a job, through increases in self-esteem, socialization, opportunities to use skills and abilities, external structure, and income. Supported employment plans, such as Individualized Placement and Support (IPS), help to place and support people with SMIs in jobs available in their community. However, people with SMIs often have difficulties keeping jobs. Research suggests these difficulties are due to cognitive deficits-underlying patterns of thought. This study will test two versions of IPS to see which produces the best outcomes for people with SMIs looking for jobs: one version will be supplemented with cognitive training (CT), which will address cognitive deficits related to work, and the other version will be supplemented with enhanced support (ES), which will increase the support people with SMIs receive with their jobs.

Participation in this study will last 24 months. Participants will first undergo a baseline assessment and then will be randomly assigned to receive IPS with CT or IPS with ES. Participants in both groups will complete one IPS session and one support session-either CT or ES-each week for 12 weeks. The IPS sessions will involve working with a vocational counselor to find a job and then receiving support in training for and maintaining that job. Participants receiving CT sessions will be taught strategies to improve attention, learning and memory, and problem-solving. Participants receiving ES will receive extra sessions of vocational support. All participants will complete assessments at six times: at study entry and after 3, 6, 12, 18, and 24 months. These assessments will include interviews about life circumstances, psychiatric symptoms, and job satisfaction. The first four assessment sessions will involve additional tests-administered with a pencil and paper or on a computer-that measure thinking, learning, memory, and problem-solving abilities.

ELIGIBILITY:
Inclusion Criteria:

* Receiving psychiatric care at UCSD Outpatient Psychiatric Services
* DSM-IV diagnosis of a severe mental illness, including schizophrenia, schizoaffective disorder, bipolar disorder, or major depressive disorder
* Unemployed in the past 30 days, but stating a goal of work
* Fluency and literacy in English

Exclusion Criteria:

* Presence of dementia
* Presence of mental retardation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2008-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Weeks worked | Measured weekly for 2 years

SECONDARY OUTCOMES:
Cognition, based on the extended Measurement And Treatment Research to Improve Cognition in Schizophrenia (MATRICS) battery | Measured at baseline and after 3, 6, 12, 18, and 24 months
Functioning | Measured at baseline and after 3, 6, 12, 18, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth W. Twamley, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Outpatient Psychiatric Services, San Diego, California, United States

REFERENCES:
- [Derived] Burton CZ, Vella L, Twamley EW. Prospective memory, level of disability, and return to work in severe mental illness. Clin Neuropsychol. 2019 Apr;33(3):594-605. doi: 10.1080/13854046.2018.1436725. Epub 2018 Feb 25. PMID 29480043